CLINICAL TRIAL: NCT03851822
Title: Prevalence and Predictors of Chronic Critical Illness in Patients With Acute Respiratory Failure
Brief Title: Prevalence and Predictors of CCI in Patients With Acute Respiratory Failure (CCI)
Acronym: CCI
Status: Completed | Type: Observational
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Alessandro Marchioni, Principal Investigator, University of Modena and Reggio Emilia
Other Study IDs: UModenaReggio3
Record Dates: First submitted 2019-02-21; First posted 2019-02-22 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic Critical Illness (CCI) is a condition associated to patients surviving an acute phase of disease and respiratory failure (ARF) although remaining dependent on mechanical ventilation (MV). The prevalence and the underlying mechanisms of CCI have not been elucidated in this population.An observational prospective cohort study was undertaken at the Respiratory Intensive Care Unit (RICU) of the University Hospital of Modena (Italy) from January 2016 to January 2018. Patients mechanically ventilated with ARF in this unit were enrolled. Demographics, diagnosis, severity scores (APACHEII, SOFA, SAPSII) and clinical conditions (septic shock, infections, acute respiratory distress syndrome [ARDS]) were recorded on admission. Respiratory mechanics and inflammatory-metabolic blood parameters were recorded on admission and within the first seven days of stay. All these variables were tested as potential predictors of CCI through appropriate univariate and multivariate analysis.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years of age
* consecutively admitted to RICU due to acute respiratory failure (ARF) requiring mechanical ventilation.

Exclusion Criteria:

* refractory shock (death < 24h)
* patient goals of care not consistent with aggressive management
* end stage COPD requiring home oxygen long term therapy or home non invasive ventilation support
* presence of interstitial lung disease
* history of neuromuscular disease
* chest wall deformities
* pregnancy
* chemotherapy or radiotherapy within the past 30 days
* evidence of neurologic injury on CT scan and GCS < 8
* tracheostomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Observational cohort
Sampling Method: Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of CCI among patients admitted to Respiratory Intensive Care Unit (RICU) for Acute Respiratory Failure | 60 days from RICU admission
  The presence of CCI was defined as the need to perform tracheostomy in ICU associated with prolonged MV (the need for ventilatory support for more than 21 consecutive days for at least 6 h per day